CLINICAL TRIAL: NCT03447808
Title: Daratumumab and Ibrutinib for Symptomatic, Treatment-Naive CLL: A Phase 1b Proof-of-Concept Study
Brief Title: Daratumumab and Ibrutinib in Treating Patients With Symptomatic Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Woyach (Other)
Responsible Party: Sponsor-Investigator, Jennifer Woyach, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17143; NCI-2018-00159 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — daratumumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab, ibrutinib) (Experimental): Patients receive daratumumab IV on days 1, 8, 15, and 22 of courses 1-2, days 1 and 15 of courses 3-6, and day 1 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Beginning course 2, patients also receive ibrutinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase Ib trials studies the side effects of daratumumab and ibrutinib and how well they work in treating patients with symptomatic chronic lymphocytic leukemia. Monoclonal antibodies, such as daratumumab, may interfere with the ability of cancer cells to grow and spread. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving daratumumab and ibrutinib may work better in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety of treatment with daratumumab and ibrutinib for previously untreated chronic lymphocytic leukemia (CLL).

II. To determine the complete response rate (CR) at the post cycle 12 response assessment following treatment with daratumumab and ibrutinib for previously untreated chronic lymphocytic leukemia (CLL).

SECONDARY OBJECTIVES:

I. To characterize the activity of daratumumab and ibrutinib as measured by overall response rate (ORR), duration of response (DOR), progression-free survival (PFS), overall survival (OS), and time-to-next treatment.

TERTIARY OBJECTIVES:

I. To measure pharmacodynamic parameters in B cells including drug occupancy of BTK and B cell receptor signaling during treatment.

II. To determine the influence of this combination on T cell and natural killer (NK) cell number and function.

III. To assess for development of mutations that may confer resistance to this combination.

IV. To assess the ability of daratumumab to clear CLL in the peripheral blood and association of CD38 expression on CLL cells with response.

OUTLINE:

Patients receive daratumumab intravenously (IV) on days 1, 8, 15, and 22 of courses 1-2, days 1 and 15 of courses 3-6, and day 1 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Beginning course 2, patients also receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) meeting criteria established in the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria for the diagnosis and treatment of CLL
* Requires therapy for symptomatic CLL in the opinion of the treating physician as defined by:

  * Evidence of marrow failure as manifested by the development or worsening of anemia or thrombocytopenia (not attributable to autoimmune hemolytic anemia or thrombocytopenia)
  * Massive (>= 6 cm below the costal margin), progressive or symptomatic splenomegaly
  * Massive nodes (>= 10 cm) or progressive or symptomatic lymphadenopathy
  * Constitutional symptoms, which include any of the following:

    * Unintentional weight loss of 10% or more within 6 months
    * Significant fatigue limiting activity
    * Fevers >= 100.5 degrees Fahrenheit (F) for 2 weeks or more without evidence of infection
    * Night sweats > 1 month without evidence of infection
* No prior chemotherapy, immunotherapy, or targeted therapy for the treatment of CLL with the exception of palliative loco-regional radiotherapy and corticosteroids for symptom control
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin >= 8 g/dL
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelets >= 30,000/mm^3
* Prothrombin time (PT)/partial thromboplastin time (PTT) =< 1.5 x ULN
* Total bilirubin =<1.5 x ULN (excepting Gilbert?s syndrome)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (unless due to liver involvement)
* Serum creatinine < 2.0 mg/dL OR creatinine clearance (Cockcroft) >= 40 mL/min/1.73 m^2
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials; men must agree to not donate sperm during and after the study; for females, these restrictions apply for 1 month after the last dose of study drug; for males, these restrictions apply for 3 months after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening; women who are pregnant or breastfeeding are ineligible for this study
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* Positive hepatitis serology:

  * Hepatitis B virus (HBV): Patients with positive serology for hepatitis B defined as positivity for hepatitis B surface antigen (HBsAg) or hepatitis B virus core antibody (anti-HBc); patients who are positive for anti-HBc may be considered for inclusion in the study on a case-by-case basis if they are hepatitis B viral deoxyribonucleic acid (DNA) negative and are willing to undergo ongoing HBV DNA testing by real-time polymerase chain reaction (PCR); patients with positive serology may be referred to a hepatologist or gastroenterologist for appropriate monitoring and management

    * Patients with positive hepatitis B surface antigen (HBSAg) consistent with prior vaccination to HBV (i.e., hepatitis B virus surface antibody [anti-HBs]+, anti-HBc-) may participate
    * Patients suspected to have false positive serologic studies because of IV immunoglobulin administration are potentially eligible after negative PCR studies for viral DNA/ribonucleic acid (RNA) and discussion with the principal investigator
  * Hepatitis C virus (HCV): Patients with positive hepatitis C serology unless HCV RNA is confirmed negative and may be considered for inclusion in the study on a case-by-case basis (e.g., patients with negative viral load after HCV-specific treatment)

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy, radiotherapy, or investigational therapy within 28 days prior to entering the study or those who have not recovered from adverse events due to agents administered more than 28 days earlier; steroids for control of disease related symptoms are permitted
* Patients who are receiving any other investigational agents
* History of stroke or intracranial hemorrhage within 6 months prior to randomization
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Active Richter's transformation
* Known active involvement of the central nervous system by lymphoma or leukemia
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon); patients may be eligible if able to be taken off warfarin and started on an alternative anticoagulant
* Requires chronic treatment with strong CYP3A inhibitors
* Known infection with the human immunodeficiency virus (HIV) virus
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association functional classification
* History of severe (defined as grade 4 and/or requiring permanent discontinuation of prior antibody therapy) allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
* A female patient who is pregnant or breast-feeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second [FEV1] < 50% of predicted normal), persistent asthma, or a history of poorly controlled asthma within the last 2 years (controlled intermittent asthma or controlled mild persistent asthma is allowed)
* History of other active malignancies other than CLL within the past 3 years prior to study entry, with the exception of adequately treated in situ carcinoma or the cervix uteri or breast, basal cell or localized squamous cell carcinoma of the skin, previous malignancy confirmed and surgically resected (or treated with other modalities) with curative intent or without relapse for >= 2 years
* Vaccination with a live vaccine < 28 days prior to the start of treatment
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator?s opinion, could compromise the subject?s safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) + complete response with incomplete marrow recovery (CRi) defined by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria | Up to 2 years
Incidence of adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years
  Will be tabulated by type and grade and displayed in summary form.

SECONDARY OUTCOMES:
Duration of response (DOR) | From the date of first response until the date of progression or death presumed attributable to disease progression, whichever occurs first, assessed up to 2 years
  Will be summarized by the Kaplan-Meier method.
Overall survival | From the first treatment date until the date of death or date last known alive, assessed up to 2 years
  Will be summarized by the Kaplan-Meier method.
Overall survival (CR + CRi + partial response [PR]) | Up to 2 years
  With a 95% confidence interval (CI) will be reported for all evaluable patients, assuming a binomial distribution.
Progression-free survival | From the first treatment date until the date of progression or death, whichever occurs first, assessed up to 2 years
  Will be summarized by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Woyach, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu